CLINICAL TRIAL: NCT04312971
Title: Effects of Norepinephrine Infusion During Cardiopulmonary Bypass on Perioperative Changes in Lactic Acid Level: A Randomized Controlled Study
Brief Title: Norepinephrine Infusion During Cardiopulmonary Bypass
Acronym: Norcal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Norcal-03-2020
Record Dates: First submitted 2020-03-15; First posted 2020-03-18 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass
MeSH Terms: interventions — Norepinephrine

STUDY DESIGN:
Intervention Model Description: A single center, interventional, parallel, double-blind (patient - and outcome-assessor), prospective, trial in patients scheduled for elective cardiac procedures using CPB. The RCT will be conducted according to Good Clinical Practice (GCP) Guidelines and comply with the principles of the Declaration of Helsinki. The RCT will be registered in a public registry, and the study protocol with its statistical analysis plan will be published before enrolment of the first patient.
Who Masked: Participant, Outcomes Assessor
Masking Description: The placebo and the norepinephrine solutions look identical and their infusions will be continued until 60 min after skin closure. The test solution will be prepared by one anesthesiologist before the induction of anesthesia.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion of normal Saline 0.9%will be started following arterial cannulation before initiation of cardiopulmonary bypass and continued until aortic declamping time.
  Interventions: Drug: Placebo; Other: Increase infusion rate; Other: Decrease infusion rate
- Norepinephrine (Active Comparator): Infusion of norepinephrine (40 µg/ml) will be started following arterial cannulation before initiation of cardiopulmonary bypass and continued until aortic declamping time.
  Interventions: Drug: Norepinephrine; Other: Increase infusion rate; Other: Decrease infusion rate

INTERVENTIONS:
Drug: Placebo — Patients undergoing different cardiac surgical procedures will receive a continuous intravenous infusion of Normal Saline 0.9% with a starting dose of 0.0025 ml/kg/min.
  Arms: Placebo
Drug: Norepinephrine — Patients undergoing different cardiac surgical procedures will receive a continuous intravenous infusion of norepinephrine (40 ug/ml) with a starting dose of 0.0025 ml/kg/min.
  Arms: Norepinephrine
Other: Increase infusion rate — Infusion rate will be increased as needed in order to maintain a MAP ≥65 mmHg during cardiopulmonary bypass period as per the discretion of the anesthesiologist using 0.00125 ml/kg/min increments
Other: Decrease infusion rate — Infusion rate will be decreased as needed in order to maintain a MAP ≥65 mmHg during cardiopulmonary bypass period as per the discretion of the anesthesiologist using 0.00125 ml/kg/min decrements

SUMMARY:
The primary objective is to test the efficacy and safety of the accuracy of continuous intravenous infusion of norepinephrine during cardiopulmonary bypass (CPB) on the prevention of hyperlactatemia after cardiac surgery.

"Efficacy" would be tested with measurement of the postoperative changes in lactic acid level over time from the baseline value before induction of general anesthesia.

"safety" would be tested with observing the post-cardiotomy need for inotropic and vasopressor support, the incidence of postoperative acute kidney injury (AKI), changes in cardiac troponin level (CnTnI), and signs of ischemic splanchnic injury.

DETAILED DESCRIPTION:
Rationale

1.1. Vasoplegia and cardiac surgery:

Vasoplegia Syndrome (VS), prevailing in about 20% of cardiac surgical procedures (1), is defined as low mean arterial pressure (MAP) with normal or high cardiac indices and which is resistant to treatment with the commonly used vasopressors. (2,3) Vasoplegia might occur either during or after the cardiopulmonary bypass periods or during the postoperative period during the intensive care unit (ICU) stay. (3) Many factors have been found to be related to the increased Vasoplegia during the cardiopulmonary bypass period such as left ventricular ejection fraction more than 40%, male patients, elderly patients, higher body mass index, long cardiopulmonary bypass time, hypotension upon the start of cardiopulmonary bypass, perioperative use of angiotensin-converting enzyme inhibitors (ACE) and presence of infective endocarditis. (4,5)

1.2. Effects of Cardiopulmonary bypass (CPB) on Post cardiotomy Vasoplegia.

Cardiopulmonary bypass itself may intensify the effects of vasoplegia due to hemodilution which decreases the blood viscosity, so, reducing the overall peripheral vascular resistance. Moreover, the interaction of blood with the tubing of the cardiopulmonary bypass machine results in the release of inflammatory mediators which play an important role in reducing the peripheral resistance and aggravating the hypotension. Although compensatory and auto-regulatory mechanisms play an important role in maintaining adequate tissue perfusion, hypotension during the cardiopulmonary bypass period may result in poor outcomes as postoperative stroke (4) especially if the mean arterial pressure is below 65 mmHg. (6)

1.3. Hyperlactatemia after cardiac surgery

Lactate was used as a marker for adequate tissue perfusion since the mid-1800s. Although the literature has illustrated the undesirable effects of high lactate levels, however, the cause, the prevention as well as treatment measures of hyperlactatemia remain obscure. Additionally, lactic acidosis or hyperlactatemia might occur in cases of refractory vasoplegia. A rise in lactate levels is common during cardiac surgery and is well known for its deleterious and its association with poor patients' outcomes. (7)

Owing to its detrimental effects, measures to reduce the effects and treat vasoplegia were used. Firstly, excluding any equipment or mechanical failure such as the arterial line monitor, adjusting the bypass flows for higher cardiac index (CI>2.2), confirming the proper cannula position and ruling out any aortic dissection.

Secondly, adjusting some physiological parameters is of great value as checking hematocrit level for excessive hemodilution, adjusting the anesthetics with severe vasodilatory properties, excluding the possibility of a drug reaction or anaphylaxis and temperature management during hypothermic bypass.

Thirdly, the use of conventional vasopressor agents as phenylephrine, norepinephrine, and vasopressin. Finally, the use of some off-label agents as vitamin C, hydroxocobalamin, angiotensin 2, methylene blue and prostaglandin inhibitors. (8)

1.4. Why this clinical trial?

The use of norepinephrine during CPB has its own potential benefits. It is not clear if the use of continuous norepinephrine infusion during CPB would be effective and safe in lessening the postoperative hyperlactatemia and development of vasoplegia after cardiac surgery.

The here proposed randomized controlled clinical trial will test the use of continuous norepinephrine infusion during CPB with respect to the efficacy and safety to reduce the postoperative rise in blood lactate level.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status between ІІІ and ІV
* Scheduled for any type of elective cardiac surgery using CPB
* General anesthesia provided in an endotracheally intubated patient.

Exclusion Criteria:

* Decline consent to participate.
* Emergency surgery.
* Ejection fraction (EF%) less than 35%.
* Scheduled for re-do surgery.
* Scheduled for emergency surgery.
* Preoperative ventilator or circulatory support.
* Body mass index (BMI) greater than 40 Kg/m2.
* History of alcohol abuse.
* History of drug abuse.
* Pregnancy.
* Consent for another interventional study during anaesthesia
* No written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Changes in lactic acid level | For 24 hours after surgery from the start of surgery
  perioperative changes in lactic acid level measured from arterial or venous blood

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | For 24 hours after surgery from the start of surgery
  invasive arterial blood pressure measurement
Cardiac Index (CI) | For 24 hours after surgery from the start of surgery
  measured as l/min/m2
Systemic Vascular Resistance index (SVRI) | For 24 hours after surgery from the start of surgery
  measured as dynes.sec.m2/cm5
Stroke volume variation (SVV) | For 24 hours after surgery from the start of surgery
  measured as ml/min/m2
Need for rescue doses of phenylephrine | For the time of surgery
  Use of rescue doses of phenylephrine
Need for rescue doses of norepinephrine | For the time of surgery
  Use of rescue doses of norepinephrine
Need for rescue doses of ephedrine | For the time of surgery
  Use of rescue doses of ephedrine
Need for rescue doses of nitroglycerine | For the time of surgery
  Use of rescue doses of nitroglycerine
Need for rescue doses of labetalol | For the time of surgery
  Use of rescue doses of labetalol
Need for rescue doses of esmolol | For the time of surgery
  Use of rescue doses of esmolol
Need for rescue doses of atropine | For the time of surgery
  Use of rescue doses of atropine
Need for rescue doses of glycopyrrolate. | For the time of surgery
  Use of rescue doses of glycopyrrolate
Intraoperative hypoxemia | For the time of surgery
  Decrease of peripheral oxygen saturation less than 92%
Intraoperative hypercapnia | For the time of surgery
  Increase in end tidal carbon dioxide more than 45 mm Hg
Intraoperative hypotension | For the time of surgery
  Number of drops in systolic arterial pressure < 90 mmHg for 3 minutes or longer for any reasons
Intraoperative bradycardia | For the time of surgery
  Number of drops in heart rate lower than 40 beats.min-1 or 10% of baseline value for more than three minutes for any reasons.
Intraoperative myocardial ischemic episodes | For the time of surgery
  Remarkable ischemic changes included those patients with ≥ 1- mv ST-segment depression or ≥ 2-mv ST-segment elevation lasting more than 1 minute
Number of patients who required pacemaker insertion | For the time of surgery
  Need for pacemaker insertion following termination of cardiopulmonary bypass.
Number of patients who required direct current shocks | For the time of surgery
  Need for direct current shock following termination of cardiopulmonary bypass..
Number of patients who need for epinephrine | For the time of surgery
  Need for epinephrine following termination of cardiopulmonary bypass.
Number of patients who need for norepinephrine | For the time of surgery
  Need for norepinephrine following termination of cardiopulmonary bypass.
Number of patients who need for dobutamine | For the time of surgery
  Need for dobutamine following termination of cardiopulmonary bypass.
Number of patients who need for milrinone | For the time of surgery
  Need for milrinone following termination of cardiopulmonary bypass.
Number of patients who need for for Intra-Aortic Balloon Pump | For the time of surgery
  Need for intra-aortic balloon counter pulsation pump following termination of cardiopulmonary bypass.
Intraoperative need for blood transfusion | For the time of surgery
  The amount of transfused units of blood and blood products
Intraoperative fluid intake | For the time of surgery
  The amount of infused crystalloids and colloids
ICU Stay | For 30 days after surgery
  Length of ICU stay
Hospital Stay | For 30 days after surgery
  Length of hospital stay
Mortality at 30 days | For 30 days after surgery
  Alive or dead on postoperative day 30
Mortality at 90 days | For 90 days after surgery
  Alive or dead on postoperative day 90
Postoperative need for reintubation | For 30 days after surgery
  Postoperative need for reintubation during the first 30 days following surgery
Postoperative bleeding | For 30 days after surgery
  Postoperative bleeding during the first 30 days following surgery
Postoperative cardiogenic shock | For 30 days after surgery
  Postoperative cariogenic shock for the first 30 days following surgery
Postoperative acute kidney injury | For 30 days after surgery
  Postoperative acute kidney injury for the first 30 days following surgery
Postoperative splanchnic ischemia | For 30 days after surgery
  Postoperative mesenteric or splanchnic ischemia for the first 30 days following surgery
Postoperative myocardial ischemia | For 30 days after surgery
  Postoperative acute coronary syndrome for the first 30 days following surgery
Postoperative wound infection | For 30 days after surgery
  Postoperative wound infection for the first 30 days following surgery
Postoperative pneumonia | For 30 days after surgery
  Postoperative pneumonia for the first 30 days following surgery
Postoperative mediastinitis | For 30 days after surgery
  Postoperative mediastinitis for the first 30 days following surgery
Postoperative hypoxemia | For 30 days after surgery
  Postoperative decrease in peripheral oxygen saturation less than 90 for the first 30 days following surgery
Postoperative stroke | For 30 days after surgery
  Postoperative stroke for the first 30 days following surgery
Postoperative sternotomy | For 30 days after surgery
  Postoperatively during hospital stay
Postoperative sternal dehiscence | For 30 days after surgery
  Postoperatively during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Study Chair — College of Medicine, Imam Abdulrahman Bin Faisal University
Locations (2):
- Saudi Arabia (2):
  - Dammam University, Khobar, Eastern Province
  - Imam Abdulrahamn Bin Faisal University (Former, Dammam University), Dammam, Esatern

IPD SHARING:
Plan to Share IPD: Yes
The database will be locked as soon as all data are entered, and all discrepant or missing data are resolved - or if all efforts are employed and the investigators consider that the remaining issues cannot be fixed. At this step, the data will be reviewed before database locking. After that, the study database will be locked and exported for statistical analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study
Access Criteria: Permission for access to the database will be removed for all investigators, and the database will be archived.

REFERENCES:
- [Background] Tsiouris A, Wilson L, Haddadin AS, Yun JJ, Mangi AA. Risk assessment and outcomes of vasoplegia after cardiac surgery. Gen Thorac Cardiovasc Surg. 2017 Oct;65(10):557-565. doi: 10.1007/s11748-017-0789-6. Epub 2017 Jun 13. PMID 28612323
- [Background] Fischer GW, Levin MA. Vasoplegia during cardiac surgery: current concepts and management. Semin Thorac Cardiovasc Surg. 2010 Summer;22(2):140-4. doi: 10.1053/j.semtcvs.2010.09.007. PMID 21092891
- [Background] Shaefi S, Mittel A, Klick J, Evans A, Ivascu NS, Gutsche J, Augoustides JGT. Vasoplegia After Cardiovascular Procedures-Pathophysiology and Targeted Therapy. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):1013-1022. doi: 10.1053/j.jvca.2017.10.032. Epub 2017 Oct 27. PMID 29223724
- [Background] Truby LK, Takeda K, Farr M, Beck J, Yuzefpolskaya M, Colombo PC, Topkara VK, Mancini D, Naka Y, Takayama H. Incidence and Impact of On-Cardiopulmonary Bypass Vasoplegia During Heart Transplantation. ASAIO J. 2018 Jan/Feb;64(1):43-51. doi: 10.1097/MAT.0000000000000623. PMID 28777136
- [Background] Chan JL, Kobashigawa JA, Aintablian TL, Li Y, Perry PA, Patel JK, Kittleson MM, Czer LS, Zarrini P, Velleca A, Rush J, Arabia FA, Trento A, Esmailian F. Vasoplegia after heart transplantation: outcomes at 1 year. Interact Cardiovasc Thorac Surg. 2017 Aug 1;25(2):212-217. doi: 10.1093/icvts/ivx081. PMID 28459983
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Cotter EK, Kidd B, Flynn BC. Elevation of Intraoperative Lactate Levels During Cardiac Surgery: Is There Power in This Prognostication? J Cardiothorac Vasc Anesth. 2020 Apr;34(4):885-887. doi: 10.1053/j.jvca.2019.11.049. Epub 2019 Dec 9. No abstract available. PMID 31899137
- [Background] Ortoleva J, Shapeton A, Vanneman M, Dalia AA. Vasoplegia During Cardiopulmonary Bypass: Current Literature and Rescue Therapy Options. J Cardiothorac Vasc Anesth. 2020 Oct;34(10):2766-2775. doi: 10.1053/j.jvca.2019.12.013. Epub 2019 Dec 14. PMID 31917073